CLINICAL TRIAL: NCT01009125
Title: Randomized Trial of Financial Incentives to Increase Response Rates to a Mailed Survey of Healthcare Access and Utilization Among Living Kidney Donors
Brief Title: Healthcare Access and Utilization Among Living Kidney Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Barnabas Medical Center (Other)
Responsible Party: Francis L. Weng, MD, St. Barnabas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBMC-2009-40
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Organ Donor
Keywords: questionnaires; health care surveys/methods; motivation; living donors; living kidney donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- $2 cash incentive (Experimental)
  Interventions: Other: $2 cash
- $5 cash incentive (Experimental)
  Interventions: Other: $5 cash

INTERVENTIONS:
Other: $2 cash — $2 cash incentive will be included in the mailed survey
  Arms: $2 cash incentive
Other: $5 cash — $5 cash incentive will be included in the mailed survey
  Arms: $5 cash incentive

SUMMARY:
This is a mailed survey to persons who served as living kidney donors at Saint Barnabas Medical Center. The experimental component of this study (the clinical trial) is a randomized trial of two monetary incentives for the living kidney donors invited to participate in the study. Kidney donors will be randomized to receive one of two incentives in the mailed survey packet: $2 cash vs. $5 cash. The main outcome measure is the response rate to the survey.

ELIGIBILITY:
Inclusion Criteria:

* Persons who donated a living donor kidney at Saint Barnabas Medical Center between January 2000 and December 2006 are eligible to participate

Exclusion Criteria:

* Current address outside the continental United States
* Persons who donated a living donor kidney prior to January 2000 or after December 2006
* Persons who indicated they no longer wished to be contacted by Saint Barnabas Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Survey response rate | 2 weeks, 2 months (primary), 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Francis L Weng, MD, Principal Investigator — St. Barnabas Medical Center
Locations (1):
- Saint Barnabas Medical Center, Livingston, New Jersey, United States